CLINICAL TRIAL: NCT00895791
Title: Comparison of Healing Responses After Treatment of Complex Bifurcation Lesions With the AXXESS Biolimus A9 Eluting Stent Versus Culotte Technique Using Everolimus-eluting Stents: an Optical Coherence Tomography Analysis.
Brief Title: COmplex BifuRcation Lesions: A Comparison Between the AXXESS Device and Culotte Stenting: An Optical Coherence Tomography (OCT) Study
Acronym: COBRA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: major protocol changes: new study submitted
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Eudract: 2009-010879-24
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2009-05

CONDITIONS: Coronary Artery Stenosis
Keywords: coronary bifurcation; stent implantation; PCI; Optical Coherence Tomography
MeSH Terms: conditions — Coronary Stenosis

ARMS (2):
- 1 (Active Comparator): AXXESS Biolimus A9-eluting bifurcation stent
  Interventions: Device: AXXESS Biolimus A9-eluting bifurcation stent
- 2 (Active Comparator): culotte stenting with use of 2 drug eluting stents
  Interventions: Device: culotte stenting (Xience V)

INTERVENTIONS:
Device: AXXESS Biolimus A9-eluting bifurcation stent — implantation of stent
  Arms: 1
Device: culotte stenting (Xience V) — implantation of stent
  Other Names: culotte stenting with Xience V
  Arms: 2

SUMMARY:
The aim of this study is to compare vessel healing at 9 months using OCT imaging for two different treatment techniques for treating bifurcation lesions. Quantitative assessment of OCT images will be used to assess re-endothelialization and quality of strut apposition to the vessel wall.

DETAILED DESCRIPTION:
Background: There is an ongoing controversy over the efficacy and safety of different bifurcation stenting techniques. Critical considerations are the rate of restenosis at the side branch ostium, and completeness of healing at sites of overlap of stent struts, which may affect the risk of stent thrombosis.

Methods: Patients with complex bifurcation lesions with involvement of a significant side branch requiring a stent are randomized into two treatment arms. The first group of 20 patients (group I) is treated with the AXXESS Biolimus A9 Bifurcation Stent System (Devax, Inc, Lake Forest CA), where additional everolimus-eluting Xience V stents (Abbott Vascular, Santa Clara, CA) are implanted into the distal main branch and the side branch as required. The second group of 20 patients (group II) is treated with the culotte technique using everolimus-eluting Xience V stents. Kissing balloon dilatation using non-compliant balloons will complete the index procedure in all cases. At 9 months, control angiography (with QCA using dedicated software) and OCT (of both main vessel and side branch) is performed.

Assessment of Results:

1. EP: stent strut coverage and stent strut apposition, assessed with OCT at 9 months.
2. EP: restenosis, restenosis at SB ostium, MACE, stent thrombosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient older than 18 years
2. Written informed consent available
3. Patient eligible for percutaneous coronary intervention
4. Patients with a de novo and true coronary bifurcation lesion (Medina classification (1,1,1), (1,0,1) or (0,1,1))
5. Target reference vessel diameter measured by QCA: 2-4 mm
6. Target lesion stenosis measured by QCA: > 70% - < 100%
7. Patients willing to provide written informed consent prior to participation and willing and able to participate in all follow-up evaluations

Exclusion Criteria:

1. Left ventricular ejection fraction of < 30%
2. Impaired renal function (serum creatinine > 2.0 mg/dl)
3. Previous and/or planned brachytherapy of target vessel
4. Lesion of the left main trunk > 50%, unprotected
5. Known allergies to antiplatelet, anticoagulation therapy, contrast media or everolimus
6. Pregnant and/or breast-feeding females or females who intend to become pregnant (pregnancy test required)
7. Patients with a life expectancy of less than one year
8. Patient currently enrolled in other investigational device or drug trial
9. Patient not able or willing to adhere to follow-up visits
10. Patients who intend to have a major surgical intervention within 6 months of enrolment in the study
11. Patient not able or willing to adhere to follow-up visits
12. Patients who previously participated in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is % stent strut coverage and % stent strut apposition, assessed with optical coherence tomography, at 9 months follow-up. | 9 months

SECONDARY OUTCOMES:
Clinical outcome: Cumulative MACE rate at 1, 8, 9 and 12 months, yearly until 5 years. Separate rates will be provided for: cardiac death, non-fatal myocardial infarction, clinically driven TLR, TVR. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tom Adriaenssens, MD, Principal Investigator — UZLeuven, cardiology; Walter Desmet, MD, PhD, Study Director — UZ Leuven, Cardiology
Locations (1):
- UZ Leuven Cardiology, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided